CLINICAL TRIAL: NCT03728335
Title: Phase 2 Trial of Enasidenib (AG-221) Maintenance Post Allogeneic Hematopoietic Cell Transplantation in Patients With IDH2 Mutation
Brief Title: Enasidenib (AG-221) Maintenance Post Allogeneic HCT in Patients With IDH2 Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18117; NCI-2018-02371 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18117 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 2-Propanol; methanesulfonic acid; enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (enasidenib mesylate) (Experimental): Patients receive enasidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enasidenib Mesylate

INTERVENTIONS:
Drug: Enasidenib Mesylate — Given PO
  Other Names: 2-Methyl-1-[(4-[6-(trifluoromethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyridin-4-yl]amino}-1,3,5-triazin-2-yl)amino]propan-2-ol Methanesulfonate; 2-Propanol, 2-Methyl-1-((4-(6-(trifluoromethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triazin-2-yl)amino)-, Methanesulfonate (1:1); AG-221 Mesylate; CC-90007; Enasidenib Methanesulfonate; Idhifa

SUMMARY:
This phase II trial studies the side effects of using enasidenib as maintenance therapy in treating patients with acute myeloid leukemia with IDH2 mutation following donor stem cell transplant. Enasidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. Evaluate the efficacy of enasidenib as post-HCT maintenance therapy in patients with mIDH2 AML, at 2-years post-HCT.

SECONDARY OBJECTIVES:

1. Assess overall (OS) and leukemia-free survival (LFS) at 1 and 2 years post-HCT;
2. Estimate the cumulative incidence of chronic GVHD at 1 and 2 years post-HCT;
3. Estimate the cumulative incidence of relapse, non-relapse mortality (NRM), GVHD and relapse free survival (GRFS) at 1 and 2 years post-HCT.

EXPLORATORY OBJECTIVES:

1. Monitor disease status among subset of patients with MRD positive disease when start to receive Enasidenib by multiparameter flow cytometry post allogeneic HCT on patients BM on days +100 and +365;
2. Investigate clearance of IDH2 mutation post HCT by NGS-PCR testing on the bone marrow specimens on days +100 and +365 and in peripheral blood every 3 months till 2 year follow up; and

OUTLINE:

Patients receive enasidenib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and periodically thereafter up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) =< 2 or Karnofsky performance status (KPS) >= 70
* Recipients of allogeneic HCT - all stem cell sources including sibling, unrelated, mismatched related/unrelated, cord and haploidentical transplant patients will be included
* Conditioning regimen: Investigator's choice based on center guidelines
* GvHD prophylaxis: sirolimus + tacrolimus or tacrolimus + methotrexate or investigator choice
* Patients must have acute myeloid leukemia (AML) with IDH2 mutation at diagnosis. Day 30 marrow post HCT should show evidence of morphologic remission with < 5% bone marrow blasts. Patients with MRD either by flow cytometry or IDH2 mutation testing will be allowed
* Patients with previous therapy with IDH2 inhibitors will be included
* Absolute neutrophil count (ANC) > 1000 (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Hemoglobin >= 9.5 gm% (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelets > 50,000/mm^3 (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelets >= 20,000/mm^3 (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Patients with lower counts can enroll if infection cytomegalovirus (CMV)/human herpesvirus 6 (HHV6) etc. is being treated actively
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Total bilirubin < 2.0 mg/dl-exception permitted in patients with Gilbert's Syndrome (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferases (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x ULN, patients with abnormal liver function tests (LFTs) in the context of active GVHD will not be included (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Creatinine clearance of >= 40/min/1.73 m^2 for participants with creatinine levels above institutional normal per 24 hour urine test or the Cockcroft-Gault formula (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Corrected QT (QTc) =< 480 ms

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* Seronegative for human immunodeficiency virus (HIV) antigen/antibody (Ag/Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR])

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Active diarrhea considered clinically significant and may impair oral drug administration
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics

  * Active infection. Patients with treated viral, bacterial or fungal infections that are controlled on therapy will be allowed to participate
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Diagnosis of Gilbert's disease
* Other active malignancy. Participants with history of prior malignancy treated with curative intent who achieved complete response (CR) more than 2 years before study entry are eligible. This exclusion rule does not apply to non-melanoma skin tumors and in-situ cervical cancer
* Females only: Pregnant or breastfeeding
* Active grade II-IV acute GVHD and/or requiring systemic steroids with prednisone dose equivalent of >= 0.25 mg/kg at end of 4 weeks
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants, who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days post treatment completion
  Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

SECONDARY OUTCOMES:
Overall survival (OS) | From starting enasidenib to date of death, assessed up to 2 years
  Will be analyzed using the Kaplan-Meier curves.
Leukemia free survival (LFS) | From starting enasidenib to date of relapse or death, assessed up to 2 years
  Will be analyzed using the Kaplan-Meier curves.
Time to relapse | From starting enasidenib to date of relapse, assessed up to 2 years
  Time to relapse will be censored at the last disease assessment if patients are known to be alive and leukemia free.
Non-relapse mortality (NRM) | From starting enasidenib to date of death from other causes than relapse, assessed up to 2 years
  Will be analyzed using the curves of cumulative incidence.
Graft versus host disease (GvHD)-free relapse free survival (GRFS) | At 1 year mark of starting enasidenib
  Will be analyzed using the Kaplan-Meier curves.

OTHER OUTCOMES:
Minimal residual disease (MRD) disappearance (bone marrow [BM]) | At days 100 and 365
  Monitor disease status among subset of patients with MRD positive disease by multiparameter flow cytometry post allogeneic hematopoietic cell transplantation (HCT) on patients BM.
IDH2 mutation clearance (BM and peripheral blood) | At days 100 and 365 and up to 2 years
  Investigate clearance of IDH2 mutation post HCT by next generation sequencing-polymerase chain reaction (NGS-PCR) testing on the bone marrow specimens.
mIDH2 variant allele fraction (BM) | At days 100 and 365
  mIDH2 variant allele fraction (VAF) by droplet digital PCR (ddPCR) BEAMing technology on bone marrow specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida

REFERENCES:
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722